CLINICAL TRIAL: NCT03409237
Title: Evaluation of Coagulation Activation in Patients With Intracranial Hypertension After Treatment With Mannitol or Hypertonic Saline Solution.
Brief Title: Coagulation Activation by Hyperosmolar Agents in Intracranial Hypertension
Status: Withdrawn | Type: Observational
Why Stopped: No participant enrolled. The human resources to perform the study also due to the COBID emegency
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Other Study IDs: NMD-50/18
Record Dates: First submitted 2018-01-09; First posted 2018-01-24 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Intracranial Hypertension; Cerebral Edema
MeSH Terms: conditions — Intracranial Hypertension; Brain Edema | interventions — Mannitol; Saline Solution, Hypertonic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Mannitol 0.2-0.3 g/kg 4 times/day.
  Interventions: Drug: Mannitol
- Group 2: Hypertonic saline solution 3%. Continous infusion of 0,5 ml/kg/h. If necessary a loading dose of 2,5 ml/kg is administered.
  Interventions: Drug: Hypertonic saline solution
- Group 3: Hypertonic solution saline 4%. Continous infusion of 0,5 ml/kg/h. If necessary a loading dose of 2,5 ml/kg is administered.
  Interventions: Drug: Hypertonic saline solution
- Group 4: Hypertonic saline solution 7%. Continous infusion of 0,5 ml/kg/h. If necessary a loading dose of 2,5 ml/kg is administered.
  Interventions: Drug: Hypertonic saline solution

INTERVENTIONS:
Drug: Mannitol — Therapy is administered according to the clinical gold standard and until reaching and maintaining serum sodium levels between 145 e 155 meq/l and an osmolarity <320.
  Groups: Group 1
Drug: Hypertonic saline solution — Therapy is administered according to the clinical gold standard and until reaching and maintaining serum sodium levels between 145 e 155 meq/l and an osmolarity <320.
  Groups: Group 2; Group 3; Group 4

SUMMARY:
Osmotherapy consists in the therapeutic use of osmotically active substances with the aim of reducing the volume and therefore the intracranial pressure. It therefore represents an essential component in the clinical management of cerebral edema and intracranial hypertension, whether they are a consequence of head trauma, ischemic or hemorrhagic stroke, and neoplasm or neurosurgical procedures.

The current study aims at evaluating in vivo the effects on haemostasis parameters of hypertonic saline solutions at different concentration, as compared to mannitol, in patients with neuroradiological signs (CT / MRI) of cerebral edema / non-traumatic intracranial hypertension.

DETAILED DESCRIPTION:
Osmotherapy is commonly used in the treatment of intracranial hypertension (ICH) due to a variety of causes, including head trauma, intracranial neoplasia, infection or hemorrhage, and status epilepticus. The principle goal of osmotherapy is to shift fluid from the intracellular into the extracellular compartment using intravenous hyperosmolar agents, thereby reducing brain edema and improving cerebral perfusion pressure. Although 10-20% mannitol is considered the gold standard hyperosmolar agent in the treatment of ICH, mannitol-induced osmotic diuresis may cause hypovolemia and reduction in cerebral perfusion pressure. In recent years, 3.0-7.5% hypertonic saline (HTS) has gained popularity in the treatment of ICH as it has less pronounced diuretic effects and therefore does not cause hypovolemia. Indeed, in the face of hypovolemic shock and traumatic brain injury, HTS provides the advantage of volume expansion, restoring adequate cerebral perfusion pressures, and reducing brain edema, which makes it superior to mannitol in trauma patients with shock.

Both mannitol and HTS have been shown to interfere with whole blood coagulation and platelet function. This is in part due to dilutional coagulopathy. Furthermore, 7.2% HTS may directly disturb both fibrin formation and platelet function, and mannitol may interfere with coagulation by reducing clot strength. In addition, hyperosmolarity is supposed to lead to impairment of both whole blood coagulation and platelet function . In consequence, the safety of using these agents in patients with ICH and intracranial hemorrhage remains unclear. Previous in vitro studies in humans have demonstrated anticoagulant effects of both mannitol and HTS, although one clinical study failed to demonstrate any negative effect on hemostasis using either solution in patients undergoing elective intracranial surgery. However, in vivo studies in a clinical setting are lacking.

ELIGIBILITY:
Inclusion Criteria:

* Indication to osmotic therapy for cerebral edema / non-traumatic intracranial hypertension
* Age 18 - 80 years
* Body temperature between 35.5 ° C and 37.5 °C

Exclusion Criteria:

* Congenital or acquired disorders of hemostasis
* Clinical history of abnormal bleeding
* Hematologic or Renal diseases (acute or chronic renal failure II-III stage)
* Chronic or recent therapy with antiplatelet and/or anticoagulants
* Taking corticosteroids or nonsteroidal anti-inflammatory drugs (less than 4 weeks)
* Administration of macromolecular vascular filling solutions (less than 4 weeks)
* History of recent venous / arterial thromboembolic disease (less than three months)
* Moderate-severe liver dysfunction
* Anemia (hb <10 mg/dl)
* Recent transfusions (less than three months)
* Hyponatremia (Na <135 meq/l)
* Hypernatremia (Na> 155 meq/l)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (men and women) with cerebral edema / intracranial hypertension (CT / MRI neuroradiological diagnosis) on a non-traumatic basis with indication to osmotic therapy, treated on the basis of clinical and radiological evidence according to current treatment standards and meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-03 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in coagulation parameters | Before osmotic therapy (time 0), after 12 hrs infusion (time 1)
  Coagulation parameters such as thrombin and prothrombin time, fibrinogen, thrombin generation time will be measured in plasma by ELISA test or on whole blood by thromboelastography

SECONDARY OUTCOMES:
Changes in inflammation markers | Before osmotic therapy (time 0), after 12 hrs infusion (time 1)
  Inflammation markers such as C reactive protein, interleukin 6, P-selectin. E-selectin will be measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, PhD, Study Chair — IRCCS Neuromed; Fulvio Aloj, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS INM Neuromed, Department of Epidemiology and Prevention, Pozzilli, IS, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre-Healy A, Marko NF, Weil RJ. Hyperosmolar therapy for intracranial hypertension. Neurocrit Care. 2012 Aug;17(1):117-30. doi: 10.1007/s12028-011-9649-x. PMID 22090171
- [Background] Ropper AH. Hyperosmolar therapy for raised intracranial pressure. N Engl J Med. 2012 Aug 23;367(8):746-52. doi: 10.1056/NEJMct1206321. No abstract available. PMID 22913684
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. II. Hyperosmolar therapy. J Neurotrauma. 2007;24 Suppl 1:S14-20. doi: 10.1089/neu.2007.9994. No abstract available. PMID 17511539
- [Background] White H, Cook D, Venkatesh B. The use of hypertonic saline for treating intracranial hypertension after traumatic brain injury. Anesth Analg. 2006 Jun;102(6):1836-46. doi: 10.1213/01.ane.0000217208.51017.56. PMID 16717334
- [Background] Prough DS, Whitley JM, Taylor CL, Deal DD, DeWitt DS. Regional cerebral blood flow following resuscitation from hemorrhagic shock with hypertonic saline. Influence of a subdural mass. Anesthesiology. 1991 Aug;75(2):319-27. doi: 10.1097/00000542-199108000-00021. PMID 1677548
- [Background] Schmoker JD, Zhuang J, Shackford SR. Hypertonic fluid resuscitation improves cerebral oxygen delivery and reduces intracranial pressure after hemorrhagic shock. J Trauma. 1991 Dec;31(12):1607-13. doi: 10.1097/00005373-199112000-00007. PMID 1749030
- [Background] Mojtahedzadeh M, Ahmadi A, Mahmoodpoor A, Beigmohammadi MT, Abdollahi M, Khazaeipour Z, Shaki F, Kuochaki B, Hendouei N. Hypertonic saline solution reduces the oxidative stress responses in traumatic brain injury patients. J Res Med Sci. 2014 Sep;19(9):867-74. PMID 25535502
- [Background] Munar F, Ferrer AM, de Nadal M, Poca MA, Pedraza S, Sahuquillo J, Garnacho A. Cerebral hemodynamic effects of 7.2% hypertonic saline in patients with head injury and raised intracranial pressure. J Neurotrauma. 2000 Jan;17(1):41-51. doi: 10.1089/neu.2000.17.41. PMID 10674757
- [Background] Rabinovici R, Yue TL, Krausz MM, Sellers TS, Lynch KM, Feuerstein G. Hemodynamic, hematologic and eicosanoid mediated mechanisms in 7.5 percent sodium chloride treatment of uncontrolled hemorrhagic shock. Surg Gynecol Obstet. 1992 Oct;175(4):341-54. PMID 1411892
- [Background] Wilder DM, Reid TJ, Bakaltcheva IB. Hypertonic resuscitation and blood coagulation: in vitro comparison of several hypertonic solutions for their action on platelets and plasma coagulation. Thromb Res. 2002 Sep 1;107(5):255-61. doi: 10.1016/s0049-3848(02)00335-3. PMID 12479887
- [Background] Tan TS, Tan KH, Ng HP, Loh MW. The effects of hypertonic saline solution (7.5%) on coagulation and fibrinolysis: an in vitro assessment using thromboelastography. Anaesthesia. 2002 Jul;57(7):644-8. doi: 10.1046/j.1365-2044.2002.02603.x. PMID 12059821
- [Background] Reed RL 2nd, Johnston TD, Chen Y, Fischer RP. Hypertonic saline alters plasma clotting times and platelet aggregation. J Trauma. 1991 Jan;31(1):8-14. doi: 10.1097/00005373-199101000-00002. PMID 1986137
- [Background] Delano MJ, Rizoli SB, Rhind SG, Cuschieri J, Junger W, Baker AJ, Dubick MA, Hoyt DB, Bulger EM. Prehospital Resuscitation of Traumatic Hemorrhagic Shock with Hypertonic Solutions Worsens Hypocoagulation and Hyperfibrinolysis. Shock. 2015 Jul;44(1):25-31. doi: 10.1097/SHK.0000000000000368. PMID 25784523
- [Background] Ng KF, Lam CC, Chan LC. In vivo effect of haemodilution with saline on coagulation: a randomized controlled trial. Br J Anaesth. 2002 Apr;88(4):475-80. doi: 10.1093/bja/88.4.475. PMID 12066721
- [Background] Rhind SG, Crnko NT, Baker AJ, Morrison LJ, Shek PN, Scarpelini S, Rizoli SB. Prehospital resuscitation with hypertonic saline-dextran modulates inflammatory, coagulation and endothelial activation marker profiles in severe traumatic brain injured patients. J Neuroinflammation. 2010 Jan 18;7:5. doi: 10.1186/1742-2094-7-5. PMID 20082712
- [Background] Luostarinen T, Niiya T, Schramko A, Rosenberg P, Niemi T. Comparison of hypertonic saline and mannitol on whole blood coagulation in vitro assessed by thromboelastometry. Neurocrit Care. 2011 Apr;14(2):238-43. doi: 10.1007/s12028-010-9475-6. PMID 21369792
- [Background] Hanke AA, Maschler S, Schochl H, Floricke F, Gorlinger K, Zanger K, Kienbaum P. In vitro impairment of whole blood coagulation and platelet function by hypertonic saline hydroxyethyl starch. Scand J Trauma Resusc Emerg Med. 2011 Feb 10;19:12. doi: 10.1186/1757-7241-19-12. PMID 21310047
- [Background] Gatidis S, Borst O, Foller M, Lang F. Effect of osmotic shock and urea on phosphatidylserine scrambling in thrombocyte cell membranes. Am J Physiol Cell Physiol. 2010 Jul;299(1):C111-8. doi: 10.1152/ajpcell.00477.2009. Epub 2010 Mar 17. PMID 20237147